CLINICAL TRIAL: NCT05885269
Title: Comparative Efficacy of Tacrolimus 0.1% and Clobetasol Propionate 0.05% in the Treatment of Alopecia Areata
Brief Title: Comparative Efficacy of Tacrolimus and Clobetasol Propionate in Alopecia Areata
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Combined Military Hospital Abbottabad (Other)
Responsible Party: Principal Investigator, danyal sajjad, Principal investigator, Combined Military Hospital Abbottabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMHAbbottabad2021
Record Dates: First submitted 2023-05-19; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A applied Clobetasol Propionate 0.05% (Active Comparator): Patient in group-A applied clobetasol propionate 0.05% twice daily for upto 03 months.
  Interventions: Drug: Group A applied topical Clobetasol Propionate
- Group B applied topical Tacrolimus 0.1% (Active Comparator): Group-B applied topical tacrolimus 0.1% twice daily for upto 3 months.
  Interventions: Drug: Group B applied topical Tacrolimus

INTERVENTIONS:
Drug: Group A applied topical Clobetasol Propionate — Patient in group-A applied clobetasol propionate 0.05% twice daily for upto 03 months
  Arms: Group A applied Clobetasol Propionate 0.05%
Drug: Group B applied topical Tacrolimus — Group-B applied topical tacrolimus 0.1% twice daily for upto 3 months.
  Arms: Group B applied topical Tacrolimus 0.1%

SUMMARY:
Methodology: The 70 patients of age 20 to 50 years presented to the out-patient department of CMH Abbottabad suffering from alopecia areata were enrolled. The non-probability consecutive sampling technique was used. Patient in group-A applied clobetasol propionate 0.05% twice daily, whereas Group-B applied topical tacrolimus 0.1% twice daily for upto 3 months. The Patients were assessed at baseline, 4th weeks, 8th week and 12th week after treatment of each session. Hair loss was calculated from SALT score at presentation and on follow-up after 3 months. The degree of response was assessed on the basis of hair re-growth as excellent (>75% re-growth), Marked (51-75% re-growth), moderate (26-50% re-growth), or slight (≤25% re-growth). To determine statistical significance χ2-square test, taking p-value <0.05 as significant, was used.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 20 to 50 years
* Both male and female
* Duration of illness less than 2 months
* those who never received any treatment before

Exclusion Criteria:

* Patients having duration of alopecia greater than 2 months
* Atypical alopecia areata i.e., Alopecia universalis etc
* Hypersensitivity history to topical corticosteroids or tacrolimus
* patients taking any systemic immune suppression
* pregnancy/lactation

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
The degree of response was assessed on The basis of hair regrowth as excellent, marked, moderate or slight. | 6 months
  The degree of response was assessed on the basis of hair regrowth as excellent (>75% regrowth), marked (51-75% regrowth), moderate (26-50% regrowth), or slight (≤25% regrowth)

CONTACTS AND LOCATIONS:
Locations (1):
- Danyal Sajjad, Abbottabad, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No